CLINICAL TRIAL: NCT05269862
Title: Remote Optimization, Adjustment and Measurement for Deep Brain Stimulation
Acronym: ROAM-DBS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABT-CIP-10413
Record Dates: First submitted 2022-01-17; First posted 2022-03-08 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Parkinson Disease
Keywords: ABT-CIP-10413; Virtual Clinic; Infinity DBS system
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- In-Clinic Cohort (Experimental): Subjects who are implanted with Abbott Infinity DBS systems with the Neuosphere Virtual Clinic feature, and receive programming for their DBS system in-clinic only.
  Interventions: Device: Abbott Infinity DBS systems with the NeuroSphere Virtual Clinic feature
- Virtual Clinic Cohort (Active Comparator): Subjects who are implanted with Abbott Infinity DBS systems with the Neuosphere Virtual Clinic feature, and receive programming for their DBS system with Virtual Clinic and in-clinic sessions.
  Interventions: Device: Abbott Infinity DBS systems with the NeuroSphere Virtual Clinic feature (virtual clinic and in-clinic sessions)

INTERVENTIONS:
Device: Abbott Infinity DBS systems with the NeuroSphere Virtual Clinic feature — Implant and initial programming of the Infinity DBS system for this cohort are conducted according to the sites standard of care. After initial programming, all follow-up programming for the first 3 months is conducted in-clinic (not using the Virtual Clinic feature).
  Arms: In-Clinic Cohort
Device: Abbott Infinity DBS systems with the NeuroSphere Virtual Clinic feature (virtual clinic and in-clinic sessions) — Implant and initial programming of the Infinity DBS system for this cohort are conducted according to the sites standard of care. After initial programming, all follow-up programming for the first 3 months is conducted using Virtual Clinic or in-clinic as appropriate.
  Arms: Virtual Clinic Cohort

SUMMARY:
The purpose of the ROAM-DBS study is to compare the time needed to achieve a 1 point improvement Patient's Global Impression of change (PGIC) relative to the subject's status at the end of the ADROIT initial programming visit in subjects who receive programming updates via in-clinic sessions and subjects who additionally have the option of receiving programming updates via Virtual Clinic sessions. The study intends to demonstrate shorter times to achieve benefit in the Virtual Clinic cohort.

DETAILED DESCRIPTION:
The ROAM-DBS study is a prospective, multi-center, randomized control, open-label, post-market cohort study intended to gather clinical data on the effect of the NeuroSphere Virtual Clinic feature (remote care) on the time needed to optimize DBS stimulation parameters after implant. The study will enroll up to 100 subjects from up to 15 centers in geographies where Abbott DBS systems with the Virtual Clinic feature are approved, which may include North America, and Europe. Subjects should be participants in the ADROIT study (NCT04071847). Subjects will be followed to a 3 month visit where the primary endpoint will be assessed. Subjects will be further followed for 1 year for final data assessment. Subjects will remain enrolled in ADROIT after the end of the ROAM study, and will complete the ADROIT 6 month and 1 year visits under that protocol. The study is expected to enroll subjects for up to 2 years, and complete all follow-up visits within 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a participant in the ADROIT study.
2. Subject is over 21 years old.
3. Subject is able to read and write.
4. Subject is indicated for implant with an Infinity IPG for Parkinson's disease.
5. Subject has not previously been implanted with a DBS system.
6. The treating physician believes Virtual Clinic is appropriate as a component in the treatment regime for this subject.
7. Subject will have access to the Abbott Virtual Clinic system through a participating site.
8. Subject will have internet access on their Patient Controller in a location suitable for a Virtual Clinic session.
9. Subject, or a legally acceptable representative, must provide written informed consent prior to any study-related procedure.

Exclusion Criteria:

1. Subject is currently enrolled or plans to enroll in an investigational study that may confound the results of this study.
2. Subject has anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the study or to comply with follow-up requirements, or impact the scientific soundness of the study results.
3. As assessed by the treating physician, lead misplacement would prevent the DBS therapy from providing clinically meaningful benefit.
4. Subject is unable to use the Virtual Clinic feature.
5. Subject will not be able, in the investigator's opinion, to demonstrate or articulate symptoms during a Virtual Clinic visit.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03-24 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint: The time to achieve a 1 point improvement Patient's Global Impression of change (PGIC) relative to the subject's status at the end of the initial programming visit | PGIC will be collected within 2 days (48 hours) after completion of each programming visit
  The PGI consists of 2 subscales, the first rating the severity of illness (PGIS) and the second evaluating the change in illness relative to a previous status (PGIC). The PGI scale evaluates all aspects of health and assesses if there has been a change in clinical status. The scale consists of two items, one scale rating severity of illness and one rating global improvement. Severity is rated from 1=normal/not at all ill to 7= extremely ill. Global improvement is rated from 1=very much improved to 7=very much worse. The questionnaire takes approximately 5 minutes to complete. The time needed to achieve a 1 point improvement Patient's Global Impression of change (PGIC) relative to the subject's status at the end of the initial programming visit in subjects who receive programming updates via in-clinic sessions and subjects who additionally have the option of receiving programming updates via Virtual Clinic sessions, will be compared.
Primary Safety Endpoint: Rate of programming related adverse events for the Virtual Clinic cohort | At 3-months after initial programming visit
  The rate of programming related adverse events reported up to the Short Term (3 month) follow-up visit for the Virtual Clinic cohort will be summarized using counts and percentages.

SECONDARY OUTCOMES:
Patient Global Impression (PGI) | At 3-months after initial programming visit
  The PGI consists of 2 subscales, the first rating the severity of illness (PGIS) and the second evaluating the change in illness relative to a previous status (PGIC). The PGI scale evaluates all aspects of health and assesses if there has been an improvement or decline in clinical status. The scale consists of two items, one scale rating severity of illness and one rating global improvement. Severity is rated from 1=normal/not at all ill to 7= extremely ill. Global improvement is rated from 1=very much improved to 7=very much worse. The clinical scores of virtual Clinic cohort will be compared to the in-clinic cohort.
Patient Global Impression (PGI) | At 1 Year after initial programming visit
  The PGI consists of 2 subscales, the first rating the severity of illness (PGIS) and the second evaluating the change in illness relative to a previous status (PGIC). The PGI scale evaluates all aspects of health and assesses if there has been an improvement or decline in clinical status. The scale consists of two items, one scale rating severity of illness and one rating global improvement. Severity is rated from 1=normal/not at all ill to 7= extremely ill. Global improvement is rated from 1=very much improved to 7=very much worse. The clinical scores of virtual Clinic cohort will be compared to the in-clinic cohort.
Clinical Global Impression (CGI) | At 3-months after initial programming visit
  The CGI questionnaire is widely used for assessing symptoms and consists of two subscales, one rating severity of illness (CGIS) and one rating global improvement (CGIC) (12-14). Severity is rated from 1 = normal/not at all ill to 7 = among the most extremely ill. Global improvement is rated from 1 = very much improved to 7 = very much worse. The clinical scores of virtual Clinic cohort will be compared to the in-clinic cohort.
Clinical Global Impression (CGI) | At 1 Year after initial programming visit
  The CGI questionnaire is widely used for assessing symptoms and consists of two subscales, one rating severity of illness (CGIS) and one rating global improvement (CGIC) (12-14). Severity is rated from 1 = normal/not at all ill to 7 = among the most extremely ill. Global improvement is rated from 1 = very much improved to 7 = very much worse. The clinical scores of virtual Clinic cohort will be compared to the in-clinic cohort.
Parkinson's Disease Questionnaire (PDQ-39) | At 3-months after initial programming visit
  PDQ-39 questionnaire is a widely used validated questionnaire to measure PD-specific health status (16-17). The self-administered questionnaire consists of 39 questions and assesses how often the subject has experienced difficulties during the past month due to PD across 8 dimensions including mobility, activities of daily living, emotional well-being, social support, cognition, communication and bodily discomfort. Each question is rated on a 5-point ordinal scoring system ranging from 0=never to 4=always. Each dimension total score ranges from 0 (never have difficulty) to 100 (always have difficulty). The overall score is expressed by a Summary Index. Lower scores reflect better quality of life. The clinical scores of virtual Clinic cohort will be compared to the in-clinic cohort.
Parkinson's Disease Questionnaire (PDQ-39) | At 1 Year after initial programming visit
  PDQ-39 questionnaire is a widely used validated questionnaire to measure PD-specific health status (16-17). The self-administered questionnaire consists of 39 questions and assesses how often the subject has experienced difficulties during the past month due to PD across 8 dimensions including mobility, activities of daily living, emotional well-being, social support, cognition, communication and bodily discomfort. Each question is rated on a 5-point ordinal scoring system ranging from 0=never to 4=always. Each dimension total score ranges from 0 (never have difficulty) to 100 (always have difficulty). The overall score is expressed by a Summary Index. Lower scores reflect better quality of life. The clinical scores of virtual Clinic cohort will be compared to the in-clinic cohort.
Levodopa Equivalent Dose (LED) | At 3-months after initial programming visit
  LED will be assessed and the values of virtual Clinic cohort will be compared to that of in-clinic cohort.
Levodopa Equivalent Dose (LED) | At 1 Year after initial programming visit
  LED will be assessed and the values of virtual Clinic cohort will be compared to that of in-clinic cohort.
Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | At 1 Year after initial programming visit
  MDS-UPDRS questionnaire is a widely used validated questionnaire to assess the severity of Parkinson's disease. This questionnaire is composed of four sections, however, this study shall only utilize part III: motor examinations consisting of 33 scores based on 18 questions with several right, left or other body distribution scores. Each item is scored from 0 to 4, where 0 indicates normal, 1 indicates slight symptoms, 2 indicates mild symptoms, 3 indicates moderate symptoms, and 4 indicates severe symptoms. The total score is obtained from the sum of the corresponding item scores. Higher scores indicate greater impact of PD symptoms. The clinical scores of virtual Clinic cohort will be compared to the in-clinic cohort.
Home Monitoring (Tremor) | At 3-months after initial programming visit
  Subjects will be provided with a home monitoring kit consisting of a smart watch and smart phone and will be instructed on how to use and charge the devices in order to monitor the prevalence and severity of tremor during activities of daily living. The supplied smart phone will also provide a diary function that subjects will use to maintain notes on symptoms and medications. The smart watch data provides time stamped data indicating the presence of tremor, and its severity (slight (< 0.1 cm), mild (0.1-0.6 cm), moderate (0.6-2.2 cm),strong (>2.2 cm) and absent during each one-minute interval). The Home Monitoring equipment is validated against physician assessments of tremor. Home Monitoring data is uploaded and stored in a secured cloud server.
Home Monitoring (Dyskinesia) | At 3-months after initial programming visit
  Subjects will be provided with a home monitoring kit consisting of a smart watch and smart phone and will be instructed on how to use and charge the devices in order to monitor the prevalence and severity of dyskinesia during activities of daily living. The supplied smart phone will also provide a diary function that subjects will use to maintain notes on symptoms and medications. The smart watch data provides the % of time in each 15 minute interval the subject experiences dyskinesia. The Home Monitoring equipment is validated against physician assessments of dyskinesia. Home Monitoring data is uploaded and stored in a secured cloud server.
"On Time" (time each day without troublesome symptoms or side effects) (derived from Home Monitoring) | At 3-months after initial programming visit
  "On Time" (time each day without troublesome symptoms or side effects) will be assessed by summing the daily intervals where Home Monitoring data does not measure tremor or dyskinesia
Health care resource utilization: Number of hospitalizations and ER visits | At 1 Year after initial programming visit
  The number of hospitalizations and ER visits will be assessed
Time to resolve programming related adverse events | At 1 Year after initial programming visit
  Time to resolve programming related adverse events will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Bradley White, Study Chair — Abbott; Devyani Nanduri, Study Director — Abbott Medical Devices Neuromodulation
Locations (18):
- United States (11):
  - University of Arizona Health Sciences Center, Tucson, Arizona
  - University of California at Davis, Sacramento, California
  - University of Miami Hospital, Miami, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State Medical, Columbus, Ohio
  - Thomas Jefferson Department of Neurosurgery, Philadelphia, Pennsylvania
  - Texas Movement Disorder Specialist, Georgetown, Texas
- Germany (3):
  - Universitäts Klinikum Tübingen, Tübingen, Bad-wur
  - Medizinische Einrichtungen der Universität Düsseldorf, Düsseldorf, N. RHIN
  - UNIVERSITATSMEDIZIN der Johannes Gutenberg-Universität Mainz, Mainz, Rhinela
- Spain (3):
  - Hospital Universitari Germans Trias I Pujol, Badalona
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Virgen de Rocio, Seville
- Queen Elizabeth University Hospital, Glasgow, Wdbtshr, United Kingdom

IPD SHARING:
Plan to Share IPD: No